CLINICAL TRIAL: NCT05670392
Title: The Advantage of Combined Non-ablative Erbium Yttrium Aluminum Garnet Laser and High Intensity Tesla Magnetic Stimulation for Treatment of Female Stress Urinary Incontinence
Brief Title: Laser and High Intensity Tesla Magnetic Stimulation (HITS) for Stress Urinary Incontinence (SUI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cork University Maternity Hospital (Other)
Collaborators: Fotona d.o.o. (Industry)
Responsible Party: Principal Investigator, Barry O'Reilly, Head of Urogynecology department, Cork University Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LASERHITS
Record Dates: First submitted 2022-12-20; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Stress Urinary Incontinence
Keywords: SUI; Incontinence; Laser; High Intensity Tesla Magnetic Stimulation
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: a two-arm parallel assignment, randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: laser and HITS treatment (Active Comparator): Laser and magnetic chair Treatment
  Interventions: Device: laser and High intensity Tesla magnetic stimulation
- Arm 2: laser (without HITS treatment) (Other): Laser treatment
  Interventions: Device: laser (without HITS treatment)

INTERVENTIONS:
Device: laser and High intensity Tesla magnetic stimulation — Three (3) non-ablative Er:YAG laser treatments will be applied at monthly intervals followed by Eight (8) HITS therapies) Patients will receive two (2) HITS treatments per week for four (4) weeks(.
  Arms: Arm 1: laser and HITS treatment
Device: laser (without HITS treatment) — Three (3) non-ablative Er:YAG laser treatments will be applied at monthly intervals as described above.
  Arms: Arm 2: laser (without HITS treatment)

SUMMARY:
To investigate the efficacy of combined laser and HITS treatment for female stress urinary incontinence (SUI)

DETAILED DESCRIPTION:
This study is a single-centre, two-arm randomized control trial study conducted according to Helsinki Declaration. Women with symptoms of stress urinary incontinence (SUI) (stress or mixed with stress incontinence as the predominant symptom) will be enrolled.

The efficacy and safety of combined treatment with non-ablative intravaginal Er:YAG laser procedure and high intensity Tesla magnetic stimulation will be compared to the treatment of non-ablative intravaginal Er:YAG laser alone.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female, 18 years of age or older
2. Clinical diagnosis of stress or mixed urinary incontinence, with stress incontinence as the predominant symptom (SUI or MUI)

Exclusion Criteria:

1. Very severe urinary incontinence (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) ICIQ-UI )score at baseline >18 or Pad test > 50 gr)
2. Pregnancy
3. BMI>35
4. Acute urinary tract infections (UTIs)
5. History of a genital fistula, a thin recto-vaginal septum as determined by the investigator or history of a fourth-degree laceration during screening physical exam (e.g., perineal body)
6. Active sexually transmitted disease upon vaginal exam (as determined by the investigator) that precludes treatment or any other vaginal infection
7. Prolapse grade 2 or higher
8. History of radiotherapy for cervical or uterine cancer
9. Medical condition that may interfere with participants' compliance to the protocol
10. Medical condition for which the HITS and laser therapy are contraindicated
11. Previous laser or HITS treatment for SUI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female genitalia
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms of stress urinary incontinence | measured at 3 and 6 months
  Change of symptoms of stress and/or mixed urinary incontinence as measured by change in one hour pad test (gr/h) results at the end of treatment period from the baseline results.
Adverse events | up to 6 month post procedure
  The number and severity of treatment-related Adverse Events.

SECONDARY OUTCOMES:
QUID - Questionnaire for Urinary Incontinence Diagnosis | measured at 3 and 6 months
  The Questionnaire for Urinary Incontinence Diagnosis (QUID) identifies the presence and frequency of stress and urge incontinence symptoms. Three items focus on stress incontinence symptoms and three on urge incontinence symptoms. Each item includes 6 frequency-based response options, ranging from "none of the time" to "all of the time", which are scored from 0 to 5 points. Scores are calculated in an additive fashion, resulting in separate Stress and Urge scores, each ranging from 0 to 15 points.
FSFI - The Female Sexual Function Index | measured at 3 and 6 months
  FSFI - The Female Sexual Function Index is a generalized questionnaire utilized to assess sexual function in women in a general population. It has been validated on clinically diagnosed samples of women with female sexual arousal disorder, female orgasmic disorder, and hypoactive sexual desire disorder.
  Scoring is between 2 (low sexual function)-36 (high sexual function).
PGI-I - Patient Global Impression of Improvement | measured at 3 and 6 months
  The Patient Global Impression of Improvement (PGI-I) is a global index that may be used to rate the response of a condition to a therapy (transition scale). It is a simple, direct, easy to use scale that is intuitively understandable to clinicians.
  1-7: Very much better- 1, Much better -2, A little better-3, No change-4, A little worse-5, Much worse-6, Very much worse-7.
One-hour pad test. | measured at 3 and 6 months
  he testing protocol has been standardized by International Continence Society (ICS-pad test):
  * the test is started by putting one pre-weighted pad without patient voiding,
  * patient drinks 500 ml of sodium-free liquid in <15 min- then sits or rests,
  * patient walks for 30 min, including climbing one flight of stairs (up and down),
  * patient performs the following activities: standing up from sitting (10x), coughing vigorously (10x), running on the spot for 1 min, bending to pick up an object from the floor (5x), and washing hands in running water for 1min (this activity program may be modified according to the patient's physical fitness),
  * the total amount of urine leaked is determined by weighing the pad. If a moderately full bladder cannot be maintained through the hour (if the patient must void), the test has to be started again.
International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | measured at 3 and 6 months
  The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. This short and simple questionnaire is also of use to general practitioners and clinicians in both primary and secondary care institutions to screen for incontinence, to obtain a brief yet comprehensive summary of the level, impact and perceived cause of symptoms of incontinence and to facilitate patient-clinician discussions. Scoring is between 0 to 21 (worse symptoms )

CONTACTS AND LOCATIONS:
Overall Officials: Barry O'Reilly, Prof., Principal Investigator — Cork University Maternity Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuszka A, Gamper M, Walser C, Kociszewski J, Viereck V. Erbium:YAG laser treatment of female stress urinary incontinence: midterm data. Int Urogynecol J. 2020 Sep;31(9):1859-1866. doi: 10.1007/s00192-019-04148-9. Epub 2019 Dec 11. PMID 31828400
- [Background] Chandi DD, Groenendijk PM, Venema PL. Functional extracorporeal magnetic stimulation as a treatment for female urinary incontinence: 'the chair'. BJU Int. 2004 Mar;93(4):539-42. doi: 10.1111/j.1464-410x.2003.04659.x. PMID 15008725
- [Result] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Result] He Q, Xiao K, Peng L, Lai J, Li H, Luo D, Wang K. An Effective Meta-analysis of Magnetic Stimulation Therapy for Urinary Incontinence. Sci Rep. 2019 Jun 24;9(1):9077. doi: 10.1038/s41598-019-45330-9. PMID 31235706